CLINICAL TRIAL: NCT06707129
Title: Establishment of Precise Histological Evaluation Criteria for Reversal of NASH Fibrosis
Brief Title: Establishment of Precise Histological Evaluation Criteria for NASH Fibrosis Reversal
Status: Recruiting | Type: Observational
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Minghui Li, Director and Professor of Hepatology Department 2, Beijing Ditan Hospital
Other Study IDs: ZLRK202301
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease; nonalcoholic steatohepatitis; liver biopsy; Fibrosis reversal; histopathology
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: After successful patient screening and enrollment, visits will be conducted every 6 months to collect the following information: Physical examination, accompanying diseases, hematology: blood routine, coagulation function, serology, imaging, body fat measurement, liver puncture information (if applicable). Lifestyle questionnaire: Dietary characteristics, sleep/wake time, daily sitting time, exercise duration, exercise mode. Health education and lifestyle intervention guidance should be provided to patients based on exercise mode. When adjusting lifestyle for at least 1 year and no more than 3 years, a second liver biopsy should be performed to evaluate liver histological changes.
  Interventions: Other: life-style

INTERVENTIONS:
Other: life-style — The patients were given health education and lifestyle intervention guidance, followed by lifestyle adjustment for at least 1 year and no more than 3 years, and a second liver biopsy was performed to evaluate liver histological changes.

SUMMARY:
Collect confirmed cases of NAFLD patients and enroll them in the study. Select patients with NASH and fibrosis stage F2-4 confirmed by liver biopsy, and collect clinical and pathological data for relevant evaluation and definition. Establish a NASH "fibrosis reversal" pathological evaluation system, based on a new reversal standard, establish non-invasive alternative indicators, and observe indicators.

DETAILED DESCRIPTION:
Confirmed NAFLD patients were enrolled, and those with NASH and fibrosis F2-4 stages confirmed by liver biopsy were selected, and clinical and pathological data were collected for relevant evaluation and definition. A NASH "fibrosis reversal" pathological evaluation system was established based on the new standard, and an alternative non-invasive indicator and observation index were established based on the reversal standard.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years at the time of liver biopsy;
* Gender is not limited;
* Hepatic perforation suggested that NASH complicated with fibrosis stage F2-4;
* Signed written informed consent.

Exclusion Criteria:

* Combined HCV infection, HIV infection, alcoholic liver disease, autoimmune liver disease, genetic metabolic liver disease Disease, drug-induced liver injury and other chronic liver diseases;
* Women during pregnancy;
* There are the following conditions before liver perforation: HCC or possible HCC (imaging suggests malignant liver occupation); decompensation of cirrhosis (ascites, hepatic encephalopathy, gastrointestinal bleeding, hepatorenal syndrome, etc.); Patients with other malignant tumors; Recipients of liver transplantation;
* Patients considered by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NAFLD were enrolled, and patients with NASH and fibrosis stage F2-4 confirmed by liver biopsy were screened
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Reversal of NASH liver fibrosis | 12 months
  Reversal of NASH liver fibrosis based on liver biopsy definition

SECONDARY OUTCOMES:
Changes in LSM value | 12 months
  Changes in liver stiffness value (LSM value) detected by instantaneous liver elasticity testing
Changes in liver fat content | 12 months
  Instantaneous liver elasticity detection of changes in liver fat content (CAP value)
The dynamic changes of existing non-invasive evaluation models for fibrosis | 12 months
  The dynamic changes of existing non-invasive evaluation models for fibrosis include: APRI=AST(ULN)/PLT(10^9/L)×100
The dynamic changes of existing non-invasive evaluation models for fibrosis | 12 months
  The dynamic changes of existing non-invasive evaluation models for fibrosis include:
  FIB-4: Age, AST, ALT, platelets
The dynamic changes of existing non-invasive evaluation models for fibrosis | 12 months
  The dynamic changes of existing non-invasive evaluation models for fibrosis include:
  BARD：BMI ≥28, AST/ALT ≥0.8, diabetes
The dynamic changes of existing non-invasive evaluation models for fibrosis | 12 months
  The dynamic changes of existing non-invasive evaluation models for fibrosis include:
  NAFLD Fibrosis Score
The dynamic changes of existing non-invasive evaluation models for fibrosis | 12 months
  The dynamic changes of existing non-invasive evaluation models for fibrosis include:
  FAST
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including BMI;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including body fat percentage;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including blood pressure;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including sugar;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including glycated hemoglobin;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including fasting insulin;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including uric acid;
Dynamic changes in metabolic indicators of NAFLD | 12 months
  Dynamic changes in metabolic indicators of NAFLD, including blood lipid series;
The occurrence of cirrhosis | 12 months
  The occurrence of cirrhosis: that is, when the liver biopsy did not indicate cirrhosis at the time of enrollment, cirrhosis occurred during follow-up.
The occurrence of liver outcome events | 12 months
  The occurrence of liver outcome events: decompensation of cirrhosis (ascites, rupture of esophageal and gastric varices) Blood, hepatic encephalopathy, hepatocellular carcinoma, liver related deaths/liver transplantation.
Extrahepatic related events | 12 months
  Extrahepatic related events: cardiovascular and cerebrovascular events, extrahepatic malignant tumors, and newly developed metabolic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China